CLINICAL TRIAL: NCT04598035
Title: Epidural Spinal Cord Stimulation for Hypertension in Patients With Neuropathic Pain
Acronym: ESCAPE
Status: Active, not recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Seth Holwerda PhD, Principal Investigator, University of Kansas Medical Center
Other Study IDs: 00145752
Record Dates: First submitted 2020-10-07; First posted 2020-10-22 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Chronic Pain; Hypertension; Implanted Stimulation Electrodes
MeSH Terms: conditions — Chronic Pain; Hypertension | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Primary Group: Patients with chronic low back pain that candidates them for surgical implant of a SCS device, and received a permanent SCS device.
  Interventions: Diagnostic Test: Diagnostic Tests
- Control Group: Patients with chronic low back pain that are candidates for a surgical implant of a SCS device and do not receive a permanent SCS device after trial leads are placed.
  Interventions: Diagnostic Test: Diagnostic Tests

INTERVENTIONS:
Diagnostic Test: Diagnostic Tests — 1. Blood and Urine laboratory tests
  2. ECG and blood pressure for cardiovascular measurements
  3. Self-report questionnaires about pain

SUMMARY:
The purpose of the ESCAPE Study is to determine the extent to which epidural spinal cord stimulation (SCS) reduces arterial blood pressure (BP) in patients which chronic low back pain and hypertension. We also aim to determine the extent to which higher baseline BP (i.e., hypertension) predicts reductions in pain following SCS implant. This is an observational study of patients undergoing an implantation of a SCS device.

DETAILED DESCRIPTION:
The broad research goal of this study is to examine the extent to which arterial blood pressure (BP) and blood markers related to hypertension and kidney function are reduced in a prospective cohort of patients undergoing implantation of an epidural spinal cord stimulator (SCS) for the purpose of managing chronic pain in the lower back and/or limbs.

Specific aims:

1. Examine the extent to which BP (primary variable), norepinephrine (marker of sympathetic nerve activity in the blood), and a vascular ultrasound scan are improved following the implant of a SCS device among patients with chronic pain and hypertension.
2. Examine the extent to which markers of kidney function in the blood [serum creatinine, glomerular filtration rate (GFR), and blood urea nitrogen (BUN)] are reduced following the implant of a SCS device among patients with chronic pain and hypertension.
3. Determine the extent to which BP predicts reductions in pain following the implant of a SCS device.

ELIGIBILITY:
* Planning to have an epidural spinal cord stimulation device implanted at KUMC
* Male or Female, age 30-89
* Low back pain for more than 3 months
* Willing to visit research lab
* Willing to undergo a blood draw and blood pressure measures
* Able to provide written informed consent

Ages: 30 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic low back pain (complex regional pain syndrome, failed back surgery syndrome)
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Blood Pressure Measurement to 1 week post-op | Baseline and 1 week post-op
  Measurements of blood pressure via arm cuff and finger cuff
Change from Baseline Blood Pressure Measurement to 4 week post-op | Baseline and 4 week post-op
  Measurements of blood pressure via arm cuff and finger cuff
Change from Baseline Blood Pressure Measurement to 8 week post-op | Baseline and 8 week post-op
  Measurements of blood pressure via arm cuff and finger cuff
Change from Baseline PainDETECT Questionnaire to 1 week post-op | Baseline and 1 week post-op.
  A battery of questionnaires is intended to understand key aspects of pain, mood, and function as quickly and efficiently as possible. The focus of these measures is on obtaining an accurate assessment of pain, while also asking about physical function, anxiety, and other associated somatic disturbances. These questionnaires will be taken prior to SCS implant (Baseline) and after SCS implant (1 week post-op, 4 weeks post-op, and 8 weeks post-op ) to assess and compare.
  Neuropathic Pain Descriptors: The Pain DETECT is a 9-item measure of sensory descriptors and spatial and temporal characteristics that has demonstrated utility in identifying central neuropathic pain.
Change from Baseline PainDETECT Questionnaire to 4 week post-op | Baseline and 4 week post-op.
  A battery of questionnaires is intended to understand key aspects of pain, mood, and function as quickly and efficiently as possible. The focus of these measures is on obtaining an accurate assessment of pain, while also asking about physical function, anxiety, and other associated somatic disturbances. These questionnaires will be taken prior to SCS implant (Baseline) and after SCS implant (1 week post-op, 4 weeks post-op, and 8 weeks post-op ) to assess and compare.
  Neuropathic Pain Descriptors: The Pain DETECT is a 9-item measure of sensory descriptors and spatial and temporal characteristics that has demonstrated utility in identifying central neuropathic pain.
Change from Baseline PainDETECT Questionnaire to 8 week post-op | Baseline and 8 week post-op.
  A battery of questionnaires is intended to understand key aspects of pain, mood, and function as quickly and efficiently as possible. The focus of these measures is on obtaining an accurate assessment of pain, while also asking about physical function, anxiety, and other associated somatic disturbances. These questionnaires will be taken prior to SCS implant (Baseline) and after SCS implant (1 week post-op, 4 weeks post-op, and 8 weeks post-op ) to assess and compare.
  Neuropathic Pain Descriptors: The Pain DETECT is a 9-item measure of sensory descriptors and spatial and temporal characteristics that has demonstrated utility in identifying central neuropathic pain.
Baseline Laboratory Tests | Baseline
  Serum creatinine, estimated glomerular filtration rate (eGFR), blood urea nitrogen (BUN), TNF-alpha, 8-Isoprostane
1 week post-op Laboratory Tests | 1 week post-op
  Serum creatinine, estimated glomerular filtration rate (eGFR), blood urea nitrogen (BUN), TNF-alpha, 8-Isoprostane
4 week post-op Laboratory Tests | 4 week post-op
  Serum creatinine, estimated glomerular filtration rate (eGFR), blood urea nitrogen (BUN), TNF-alpha, 8-Isoprostane
8 week post-op Laboratory Tests | 8 week post-op
  Serum creatinine, estimated glomerular filtration rate (eGFR), blood urea nitrogen (BUN), TNF-alpha, 8-Isoprostane

CONTACTS AND LOCATIONS:
Overall Officials: Seth W Holwerda, PhD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Clinical and Translational Science Unit (CTSU), Fairway, Kansas
  - The Marc A. Asher Comprehensive Spine Center at the Kansas University Medical Center, Kansas City, Kansas

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be available upon reasonable request